CLINICAL TRIAL: NCT04297371
Title: Early Detection of Cardiac Impairment and Prediction of Right Ventricular Hypertrophy in Patients With Connective Tissue Disease
Brief Title: Early Detection of Cardiac Impairment and Prediction of RV Hypertrophy in Patients With CTD
Acronym: EARLY-MYO-CTD
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-12-24R
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-03

CONDITIONS: Connective Tissue Diseases; Right Ventricular Hypertrophy
Keywords: Connective Tissue Diseases; Extracellular Volume; Myocardial Deformation; Cardiovascular Magnetic Resonance
MeSH Terms: conditions — Connective Tissue Diseases; Hypertrophy, Right Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CTD with RVH: The diagnosis of CTD was made based on the clinical classification criteria. The RVH patient was diagnosed by an echocardiography demonstration (later confirmed by CMR) of a hypertrophic RV (maximal end-diastole RV wall thickness >4 mm) due to CTD.
  Interventions: Diagnostic Test: CMR examination
- CTD without RVH: The diagnosis of CTD was made based on the clinical classification criteria.The subjects were enrolled as having non-RVH if their RV wall thickness was ≤ 4 mm (later confirmed by CMR).
  Interventions: Diagnostic Test: CMR examination
- Control group: The controls were healthy volunteers who have normal electrocardiographic and echocardiographic results and normal CMR findings
  Interventions: Diagnostic Test: CMR examination

INTERVENTIONS:
Diagnostic Test: CMR examination — After recruiting participants and collecting the baseline information, a CMR scan and a post-processed imaging procedure will be carried on in order to detect the cardiac impairment.

SUMMARY:
There have been reports suggesting that progressive RV failure and death in connective tissue disease (CTD) are related to right ventricular hypertrophy (RVH) and dilation, irrespective of pulmonary arterial hypertension (PAH). The investigators aim to identify cardiac markers that occur before RVH and to investigate predictors of RVH.

DETAILED DESCRIPTION:
Patients with connective tissue disease (CTD) frequently exhibit multi-organ pathophysiological and functional damage. The heart, one of the leading causes of CTD mortality, has attracted increasing attention. However, most patients with CTD present with nonspecific cardiac symptoms, normal ECG, and preserved left ventricular ejection fraction (LVEF) and therefore do not receive an early cardiac diagnosis. Pulmonary arterial hypertension (PAH), right ventricular (RV) dilatation and hypertrophy are the first and the most frequent cardiac findings. However, these are late-stage phenomena, which can eventually lead to death or right heart failure in CTD.Right ventricle abnormalities is associated with the risk of heart failure and cardiovascular death. RV dilation has long been considered a direct consequence of pulmonary arterial hypertension (PAH), but recently, physicians have observed RVH in CTD patients as well. RV dilation and RVH are not necessarily found in the same patient. The pathophysiology behind these issues is less well-understood. RVH progression continues even as CTD-associated PAH alleviates. This finding implies PAH might not be the sole index that leads to RVH. It would be interesting to explore factors that can predict the presence of RVH, which may reduce major adversecardiovascular events in patients with CTD.

Cardiovascular magnetic resonance (CMR) is able to depict myocardial characteristics from structure to tissue properties using cine and late gadolinium enhancement (LGE) sequences. Newly developed imaging studies to date include T1 mapping and T1-derived Manuscript ECV estimation.All the previous studies in CTD have been restricted to patients with advanced cardiac involvement. Together with clinical assessment and multi-imaging tests, the aim of the present study was to find markers to detect cardiac involvement before RVH presented, which could be important for guiding treatment decisions such as the timing and choice of pharmaceutical treatment. The combination of myocardial functional and tissue changes may offer further insight into the pathophysiology of CTD.

ELIGIBILITY:
Inclusion Criteria for CTD with RVH

* Age between 18-80 years old.
* Definite connective tissue diseases diagnosis.
* Echocardiography demonstration (later confirmed by CMR) of a hypertrophic RV when maximal end-diastole RV wall thickness >4 mm due to CTD

Inclusion Criteria for CTD without RVH

* Age between 18-80 years old.
* Definite connective tissue diseases diagnosis.
* Echocardiography demonstration (later confirmed by CMR) that maximal end-diastole RV wall thickness ≤4 mm

Inclusion Criteria for Control group:

* Absence of known systemic diseases
* Normal examinations
* Age between 18-80 years old.
* Providing written informed consent

Exclusion Criteria:

* Age <18 years old or >80 years old
* Documented coronary artery disease or prior angiography for coronary artery disease (>50% stenosis).
* Patients with known congenital heart disease or other systemic diseases that might induce RVH.
* Patients with standard metallic contraindications to CMR or an estimated glomerular filtration rate < 30 ml/min/1.73 m2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive subjects were prospectively enrolled into 3 cohorts between July 2014 and Nov 2016. The cohorts were divided as follows: the CTD patients with RVH, the CTD patients without RVH and the control group.
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of cardiac condition | within 2 days of CMR scan
  Compose of ventricular mass (g), volume (mL), ejection fraction (%) and strain (%) of both left and right ventricles.
Composite endpoint of quantitative fibrosis assessment | within 2 days of CMR scan
  Compose of percentage of extracellular volume (%) and positive rate of late gadolinium enhancement (%).

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital, School of Medicine, Shanghai Jiantong University
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No